CLINICAL TRIAL: NCT04211155
Title: Neural Correlates of the Shift in Social Buffering of Social Evaluative Threat in 11-14 Year Olds
Brief Title: Neural Correlates of the Shift in Social Buffering of Social Evaluative Threat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00006378
Record Dates: First submitted 2019-11-07; First posted 2019-12-26 (Actual); Results first posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Social Stress; Adolescent Behavior
MeSH Terms: conditions — Adolescent Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Primary Parent (Experimental): Participants will be randomly assigned to one of 3 conditions that differ by who is with them in the MRI scanner room: Primary Parent, Experimenter, No Social Partner.
  Interventions: Other: Questionnaires; Other: MRI
- Experimenter (Experimental): Participants will be randomly assigned to one of 3 conditions that differ by who is with them in the MRI scanner room: Primary Parent, Experimenter, No Social Partner.
  Interventions: Other: Questionnaires; Other: MRI
- No Social Partner (Experimental): Participants will be randomly assigned to one of 3 conditions that differ by who is with them in the MRI scanner room: Primary Parent, Experimenter, No Social Partner.
  Interventions: Other: Questionnaires; Other: MRI

INTERVENTIONS:
Other: Questionnaires — The participant will complete questionnaires, including ones on pubertal development and quality of relations with parents and friends.
Other: MRI — Within 2 weeks of the first study visit, the participant will return to the University where they will undergo MRI.

SUMMARY:
The purpose of this experiment is to determine the mechanisms through which parental buffering of stress physiology in response to social evaluative threat diminishes with pubertal development and whether this diminution of effectiveness extends to social buffering by peers (best friends) and/or other unfamiliar social partners (e.g., experimenters).

DETAILED DESCRIPTION:
On visit one, the participant will 1) be seen by a nurse who will complete a pubertal assessment exam, 2) complete questionnaires, including ones on pubertal development, screening for MRI safety, and quality of relations with parents and friends. The participant will also have a chance to experience a simulated MRI in order to determine whether they will be comfortable in an actual MRI.

Within 2 weeks the participant will return to the University where undergo the following protocol. Participants will be randomly assigned to one of 4 conditions that differ by who is with them in the scanner room: Primary Parent, Close Friend, Experimenter, No Social Partner. (N=50 per condition, 25 male, 25 female).

Once at the Center for Magnetic Resonance Research, participants and the individual who will be with the participant in the scanning room will undergo an MRI safety screening (the repeat of what the investigators completed over the phone). Girls will be shown to a changing room where the investigators will privately question them about any possibility of pregnancy. Participants will be shown into the scanning control room and one more safety check will be performed before they enter the scanner room and the scanner. If they are in one of the social buffering conditions, the social buffering partner will also enter the scanning room and will sit to the side of the scanner.

The scanning bed will then be moved into the barrel of the MRI machine. The participant will be wearing head phones to protect his/her hearing and to receive instructions from the control room. The participant will also be able to see two judges and hear the judges instructions when the participant is in the scanning control room. The participant will then complete a variant or the Trier Social Stress Test, a social evaluative stressor, which produces elevations in heart rate and cortisol.

When saliva is collected, the scanning bed is withdrawn from the barrel of the MRI machine and the participant will be able to see and briefly interact with the social partner while saliva is sampled for steroid collection. Once the scan is over the participant will return to a waiting area and complete additional questionnaires, provide additional saliva samples, and another urine sample.

ELIGIBILITY:
Inclusion Criteria:

* sufficient vision to complete assent and study procedures
* sufficient hearing to complete assent and study procedures
* sufficient language skills to provide verbal and written assent

Exclusion Criteria:

* Premature birth (less than 37 weeks)
* congenital and/or chromosomal disorders (e.g. cerebral palsy, FAS, mental retardation, Turner Syndrome, Down Syndrome, Fragile X)
* Autism Spectrum Disorders
* history of serious medical illness (e.g., cancer, organ transplant)
* youth taking systemic glucocorticoids
* youth taking beta-adrenergic medications
* diagnoses of psychiatric illness, seizure disorder or other neurological disorders
* contraindications for MRI (implanted medical device; presence of non-removal metal in or on the body, including piercings, orthodontic braces or certain permanent retainers)
* known pregnancy
* tattoos
* history of significant claustrophobia

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 208 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2023-06-24 (Actual); Study Completion 2023-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Gunnar, PhD, Principal Investigator — University of Minnesota; Kathleen Thomas, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Note, a fourth arm, Close Friend, was removed from the study protocol in 2021 with programmatic approval and zero enrollment, and therefore has no results to report. Delays caused by the COVID-19 pandemic required this cut in order to accomplish the study aims.
Groups:
- Primary Parent: Participants will be randomly assigned to one of 3 conditions that differ by who is with them in the MRI scanner room during the stressful task: Primary Parent, Experimenter, No Social Partner.
  In this case, participants will complete the stressor with the Primary Parent in the MRI room.
- Experimenter: Participants will be randomly assigned to one of 3 conditions that differ by who is with them in the MRI scanner room during the stressful task: Primary Parent, Experimenter, No Social Partner.
  In this case, participants will complete the stressor with the Experimenter in the MRI room.
- No Social Partner: Participants will be randomly assigned to one of 3 conditions that differ by who is with them in the MRI scanner room during the stressful task: Primary Parent, Experimenter, No Social Partner.
  In this case, participants will complete the stressor with No Social Partner in the MRI room.
Period: Overall Study
Arm/Group | Primary Parent | Experimenter | No Social Partner
Started | 72 | 64 | 72
Completed | 65 | 56 | 67
Not Completed | 7 | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- No Social Partner; Primary Parent; Experimenter: Participants will be randomly assigned to one of 4 conditions that differ by who is with them in the MRI scanner room: Primary Parent, Close Friend, Experimenter, No Social Partner.
  Questionnaires: The participant will complete questionnaires, including ones on pubertal development and quality of relations with parents and friends.
  MRI: Within 2 weeks of the first study visit, the participant will return to the University where they will undergo MRI.
- Total: Total of all reporting groups
Arm/Group | No Social Partner | Primary Parent | Experimenter | Total
Number analyzed (Participants) | 67 | 65 | 56 | 188
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 67 | 65 | 56 | 188
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.04 (1.05) | 12.95 (1) | 12.89 (1.10) | 12.96 (1.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 31 | 99
  Male | 33 | 31 | 25 | 89
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 5 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 58 | 55 | 47 | 160
  More than one race | 6 | 6 | 3 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Cortisol AUCi
Description: Area under the curve from initial (baseline) will be calculated and used in the analyses. Description = 9 saliva samples are collected during the course of the assessment. These samples are collected at (1) arrival for training purposes; T=0, (2) scan preparation; T=35 minutes, (3) entering scanner; T=55 minutes, (4) pre-TSST; T=75 minutes, (5) post-TSST; T=100 minutes, (6) pre-math alone; T=110 minutes, (7) post-math alone; T=120 minutes, (8) exiting scanner; T=130 minutes, (9) departure; T=140 minutes. Area under the curve at intercept (AUCi) is calculated using samples 2-7 with sample 2 as the intercept.
Time Frame: 2 hours, approx
Population: 188 participants were completed, with 67 Alone, 65 Parent, and 56 Experimenter. For each outcomes, all available analyzable data were included in results, sometimes resulting in lower n.
Measure: Mean (Standard Deviation); unit: (ug/dl)*minutes
Arm/Group | No Social Partner | Primary Parent | Experimenter
Number analyzed (Participants) | 65 | 61 | 55
(ug/dl)*minutes | -0.04 (0.29) | 0.02 (0.12) | -0.01 (0.06)

2. Primary Outcome: Change Heart Rate Response
Description: Heart rate will be derived from the EKG signal collected during periods of stress (social evaluation) and non-stress (no evaluation) during the course of the assessment. The variable, heart rate response, is a numeric output (reported in beats per minutes) from validated software (BIOPAC) which is calculated using a regression algorithm. The outcome measure will be reported as the difference between heart rate response during the period of stress and period of non-stress.
Time Frame: 2 hours
Population: Originally, we intended to capture heart rate date from EKG signal collected while the participant was in the MRI. During data extraction/analysis, we were unable to reliably separate out the interfering noise caused by the MRI scanner from the EKG signal. Therefore, these data are not available to be reported. Instead, we extracted data from a pulse oximeter reading on the available subset of participants, and report that data here.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Primary Parent | Experimenter | No Social Partner
Number analyzed (Participants) | 25 | 29 | 30
beats per minute | 6.09 (4.60) | 4.82 (11.07) | 4.18 (5.15)

3. Primary Outcome: Dorsal Anterior Cingulate: Task-related Brain Activity (Judged Math vs. Math Alone)
Description: The difference in fMRI BOLD signal intensity in the bilateral dorsal anterior cingulate cortex (dACC) between the social evaluative stress condition (judged math) and non-stress condition (math without judges). Mean group differences in signal intensity between the two math tasks were extracted from a brain region defined by the Harvard-Oxford brain atlas anterior cingulate cortex thresholded at 50% confidence and dorsal to the genu of the corpus callosum.
Time Frame: 2 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change in BOLD signal
Arm/Group | No Social Partner | Primary Parent | Experimenter
Number analyzed (Participants) | 53 | 48 | 50
% change in BOLD signal | 0.07369 (0.04541) | 0.09059 (0.04055) | 0.1669 (0.05167)

4. Primary Outcome: Left Anterior Insula: Task-related Brain Activity (Judged Math vs. Math Alone)
Description: The difference in fMRI BOLD signal intensity in the left anterior insula between the social evaluative stress condition (judged math) and non-stress condition (math without judges). Mean group differences in signal intensity between the two math tasks were extracted from a brain region defined by the Harvard-Oxford brain atlas left insula thresholded at 50% confidence and anterior to the region's midpoint.
Time Frame: 2 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change in BOLD signal
Arm/Group | No Social Partner | Primary Parent | Experimenter
Number analyzed (Participants) | 53 | 48 | 50
% change in BOLD signal | 0.06186 (0.02908) | 0.0807 (0.04315) | 0.1336 (0.02638)

5. Primary Outcome: Right Anterior Insula: Task-related Brain Activity (Judged Math vs. Math Alone)
Description: The difference in fMRI BOLD signal intensity in the right anterior insula between the social evaluative stress condition (judged math) and non-stress condition (math without judges). Mean group differences in signal intensity between the two math tasks were extracted from a brain region defined by the Harvard-Oxford brain atlas right insula thresholded at 50% confidence and anterior to the region's midpoint.
Time Frame: 2 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change in BOLD signal
Arm/Group | No Social Partner | Primary Parent | Experimenter
Number analyzed (Participants) | 53 | 48 | 50
% change in BOLD signal | 0.02742 (0.04186) | 0.05733 (0.03973) | 0.09256 (0.04243)

6. Primary Outcome: Ventromedial Prefrontal Cortex: Task-related Brain Activity (Judged Math vs. Math Alone)
Description: The difference in fMRI BOLD signal intensity in the bilateral ventromedial prefrontal cortex (vmPFC) between the social evaluative stress condition (judged math) and non-stress condition (math without judges). Mean group differences in signal intensity between the two math tasks were extracted from a brain region defined by the combination of Harvard-Oxford brain atlas frontal pole, frontal medial cortex, and subcallosal cortex thresholded at 50% confidence and ventral to the genu of the corpus callosum and medial to the lateral edges of the Harvard-Oxford brain atlas frontal medial cortex.
Time Frame: 2 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change in BOLD signal
Arm/Group | No Social Partner | Primary Parent | Experimenter
Number analyzed (Participants) | 53 | 48 | 50
% change in BOLD signal | 0.02742 (0.04186) | 0.05733 (0.03973) | 0.09256 (0.04243)

7. Primary Outcome: Left Dorsolateral Prefrontal Cortex: Task-related Brain Activity (Judged Math vs. Math Alone)
Description: The difference in fMRI BOLD signal intensity in the left dorsolateral prefrontal cortex (left dlPFC) between the social evaluative stress condition (judged math) and non-stress condition (math without judges). Mean group differences in signal intensity between the two math tasks were extracted from a brain region defined by the Harvard-Oxford brain atlas left middle frontal gyrus thresholded at 50% confidence.
Time Frame: 2 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change in BOLD signal
Arm/Group | No Social Partner | Primary Parent | Experimenter
Number analyzed (Participants) | 53 | 48 | 50
% change in BOLD signal | 0.11 (0.03105) | 0.08843 (0.04333) | 0.1492 (0.06621)

8. Primary Outcome: Right Dorsolateral Prefrontal Cortex: Task-related Brain Activity (Judged Math vs. Math Alone)
Description: The difference in fMRI BOLD signal intensity in the right dorsolateral prefrontal cortex (right dlPFC) between the social evaluative stress condition (judged math) and non-stress condition (math without judges). Mean group differences in signal intensity between the two math tasks were extracted from a brain region defined by the Harvard-Oxford brain atlas right middle frontal gyrus thresholded at 50% confidence.
Time Frame: 2 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change in BOLD signal
Arm/Group | No Social Partner | Primary Parent | Experimenter
Number analyzed (Participants) | 53 | 48 | 50
% change in BOLD signal | 0.05686 (0.04326) | 0.06929 (0.03735) | 0.1659 (0.04624)

9. Primary Outcome: Amygdala-vmPFC Connectivity: fMRI Functional Connectivity (Speech Prep vs. Rest)
Description: For each participant, signal intensity (unitless measure) will be measured using fMRI in the bilateral amygdala over a five-minute recording period. Signal intensity will also be measured using fMRI in the ventromedial prefrontal cortex (vmPFC) over the same period of time. A bivariate correlation will be conducted for these two data sets to determine functional connectivity, which will be reported as the r value of the correlation. This outcome measure will be reported as the mean difference in functional connectivity value (r, or correlation coefficient) for each buffering condition/group.
Time Frame: 2 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: difference in r-correlation coefficient
Arm/Group | No Social Partner | Primary Parent | Experimenter
Number analyzed (Participants) | 53 | 48 | 54
difference in r-correlation coefficient | 0.0225 (0.1774) | -0.0180 (0.1709) | 0.0131 (0.2193)

10. Primary Outcome: Amygdala-left dlPFC Connectivity: fMRI Functional Connectivity (Speech Prep vs. Rest)
Description: For each participant, signal intensity (unitless measure) will be measured using fMRI in the amygdala over a five-minute recording period. Signal intensity will also be measured using fMRI in the left dorsolateral prefrontal cortex (dlPFC) over the same period of time. A bivariate correlation will be conducted for these two data sets to determine functional connectivity, which will be reported as the r value of the correlation. This outcome measure will be reported as the mean difference in functional connectivity value (r, or correlation coefficient) for each buffering condition/group.
Time Frame: 2 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: difference in r-correlation coefficient
Arm/Group | No Social Partner | Primary Parent | Experimenter
Number analyzed (Participants) | 59 | 57 | 54
difference in r-correlation coefficient | 0.0332 (0.2236) | -0.0492 (0.1994) | -0.0263 (0.2150)

11. Primary Outcome: Amygdala-right dlPFC Connectivity: fMRI Functional Connectivity (Speech Prep vs. Rest)
Description: For each participant, signal intensity (unitless measure) will be measured using fMRI in the amygdala over a five-minute recording period. Signal intensity will also be measured using fMRI in the right dorsolateral prefrontal cortex (dlPFC) over the same period of time. A bivariate correlation will be conducted for these two data sets to determine functional connectivity, which will be reported as the r value of the correlation. This outcome measure will be reported as the mean difference in functional connectivity value (r, or correlation coefficient) for each buffering condition/group.
Time Frame: 2 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: difference in r-correlation coefficient
Arm/Group | No Social Partner | Primary Parent | Experimenter
Number analyzed (Participants) | 59 | 57 | 54
difference in r-correlation coefficient | 0.0548 (0.1983) | 0.0716 (0.2268) | 0.1069 (0.2095)

12. Primary Outcome: Hypothalamus-vmPFC Connectivity: fMRI Functional Connectivity (Speech Prep vs. Rest)
Description: For each participant, signal intensity (unitless measure) will be measured using fMRI in the hypothalamus over a five-minute recording period. Signal intensity will also be measured using fMRI in the bilateral ventromedial prefrontal cortex (vmPFC) over the same period of time. A bivariate correlation will be conducted for these two data sets to determine functional connectivity, which will be reported as the r value of the correlation. This outcome measure will be reported as the mean difference in functional connectivity value (r, or correlation coefficient) for each buffering condition/group.
Time Frame: 2 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: difference in r-correlation coefficient
Arm/Group | No Social Partner | Primary Parent | Experimenter
Number analyzed (Participants) | 59 | 57 | 54
difference in r-correlation coefficient | 0.0079 (0.1514) | 0.0424 (0.1779) | 0.0416 (0.2032)

13. Primary Outcome: Hypothalamus-left dlPFC Connectivity: fMRI Functional Connectivity (Speech vs. Rest)
Description: For each participant, signal intensity (unitless measure) will be measured using fMRI in the hypothalamus over a five-minute recording period. Signal intensity will also be measured using fMRI in the left dorsolateral prefrontal cortex (dlPFC) over the same period of time. A bivariate correlation will be conducted for these two data sets to determine functional connectivity, which will be reported as the r value of the correlation. This outcome measure will be reported as the mean difference in functional connectivity value (r, or correlation coefficient) for each buffering condition/group.
Time Frame: 2 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: difference in r-correlation coefficient
Arm/Group | No Social Partner | Primary Parent | Experimenter
Number analyzed (Participants) | 59 | 57 | 54
difference in r-correlation coefficient | 0.0269 (0.1390) | -0.0068 (0.1555) | 0.0010 (0.1571)

14. Primary Outcome: Hypothalamus-right dlPFC Connectivity: fMRI Functional Connectivity (Speech vs. Rest)
Description: For each participant, signal intensity (unitless measure) will be measured using fMRI in the hypothalamus over a five-minute recording period. Signal intensity will also be measured using fMRI in the right dorsolateral prefrontal cortex (dlPFC) over the same period of time. A bivariate correlation will be conducted for these two data sets to determine functional connectivity, which will be reported as the r value of the correlation. This outcome measure will be reported as the mean difference in functional connectivity value (r, or correlation coefficient) for each buffering condition/group.
Time Frame: 2 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: difference in r-correlation coefficient
Arm/Group | No Social Partner | Primary Parent | Experimenter
Number analyzed (Participants) | 59 | 57 | 54
difference in r-correlation coefficient | -0.0318 (0.1179) | 0.0109 (0.1585) | 0.0058 (0.1425)

15. Primary Outcome: Change in Salivary Alpha Amylase, AUCi
Description: salivary Alpha Amylase is used to index autonomic/sympathetic function. 9 saliva samples are collected during the course of the assessment. These samples are collected at (1) arrival; T=0, (2) scan preparation; T=35 minutes, (3) entering scanner; T=55 minutes, (4) pre-TSST; T=75 minutes, (5) post-TSST; T=100 minutes, (6) pre-math alone; T=110 minutes, (7) post-math alone; T=120 minutes, (8) exiting scanner; T=130 minutes, (9) departure; T=140 minutes. 4 samples (3-6) are assayed for salivary alpha amylase in micrograms per milliliter (sAA). Area under the curve at intercept (AUCi) is calculated using samples 3-6 with sample 3 as the intercept.
Time Frame: 2 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: (micrograms per milliliter) * minutes
Arm/Group | No Social Partner | Primary Parent | Experimenter
Number analyzed (Participants) | 65 | 61 | 54
(micrograms per milliliter) * minutes | 4.77 (23.26) | 6.76 (19.94) | 6.32 (41.1)

16. Secondary Outcome: Self Report of Stress
Description: Self-report of stress using a Likert-type scale with 5 levels of stress felt: (1) Not At All, (2) A Little, (3) Some, (4) A Lot, (5) A Whole Lot. Level of stress was reported for 4 points during the assessment: (1) How stressed did you feel when you first arrived at the University and we were walking into the building, (2) How stressful was the period of time when you were preparing your speech and thinking about what to say?, (3) How stressful was giving the speech?, (4) How stressful was the math with judges?. Mean Stress reactivity was calculated as the mean of (2, 3, 4) minus the value at arrival (1).
Time Frame: 2 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Social Partner | Primary Parent | Experimenter
Number analyzed (Participants) | 66 | 61 | 56
score on a scale | 1.74 (1.04) | 1.5 (1.15) | 1.81 (0.92)

17. Secondary Outcome: Peer Acceptance/Rejection
Description: Scale on the MacArthur Health and Behavior Questionnaire, Potential Covariate, 5pt Scale (1-5), High Scores Indicate Peer Acceptance
Time Frame: Parent report of child's general experience, collected over 30 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Social Partner | Primary Parent | Experimenter
Number analyzed (Participants) | 66 | 60 | 56
score on a scale | 3.55 (0.42) | 3.54 (0.41) | 3.51 (0.43)

18. Secondary Outcome: Behavioral Inhibition
Description: Scale on the MacArthur Health and Behavior Questionnaire. Potential Covariate, 3pt scale (0,1,2), high scores indicate inhibition
Time Frame: Parent report of child's general experience, collected over 30 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Social Partner | Primary Parent | Experimenter
Number analyzed (Participants) | 66 | 60 | 56
score on a scale | 0.64 (0.59) | 0.7 (0.51) | 0.69 (0.54)

19. Secondary Outcome: Internalizing Symptoms
Description: Higher Order Measure From the MacArthur Health and Behavior Questionnaire. Potential Covariate 3pt scale (0,1,2), high scores indicate Internalizing
Time Frame: Parent report of child's general experience, collected over 30 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Social Partner | Primary Parent | Experimenter
Number analyzed (Participants) | 66 | 60 | 56
score on a scale | 0.24 (0.18) | 0.24 (0.2) | 0.25 (0.2)

20. Secondary Outcome: Externalizing Symptoms
Description: Higher Order Measure From the MacArthur Health and Behavior Questionnaire. Potential Covariate 3pt scale (0,1,2), high scores indicate externalizing
Time Frame: Parent report of child's general experience, collected over 30 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Social Partner | Primary Parent | Experimenter
Number analyzed (Participants) | 66 | 60 | 56
score on a scale | 0.13 (0.11) | 0.12 (0.11) | 0.07 (0.08)

21. Secondary Outcome: Time Since Awakening
Description: Participants self-report the clock time that they woke up on the day of the assessment, and the clock time when the imaging test was done. The difference between these times was calculated and reported in hours. This is only a potential covariate for cortisol, which follows a circadian rhythm.
Time Frame: reported at the beginning of the 2 hour session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | No Social Partner | Primary Parent | Experimenter
Number analyzed (Participants) | 67 | 63 | 55
hours | 7.92 (2.03) | 8.15 (2.04) | 8.58 (1.79)

22. Secondary Outcome: Pretax Family Income. Potential Covariate
Description: Parents report on gross family income on an 11-point ordinal scale: (1) Less than $15,000, (2) $15,001 to $25,000, (3) $25,001 to $35,000, (4) $35,001 to $50,000, (5) $50,001 to $75,000, (6) $75,001 to $100,000, (7) $100,001 to $125,000, (8) $125,001 to $150,000, (9) $150,001 to $175,000, (10) $175,001 to 200,000, (11) $200,001 or more.
Time Frame: Parent report, collected over 30 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | No Social Partner | Primary Parent | Experimenter
Number analyzed (Participants) | 65 | 64 | 56
scores on a scale | 9 (2.1) | 8 (2.2) | 8 (2.1)

23. Secondary Outcome: Parental Average Education Level. Potential Covariate
Description: Parents report education level for both parents on a 6-point ordinal scale: (1) Less than high school degree, (2) High school or GED, (3) Associate degree, college academia program, (4) Bachelor's degree, (5) Master's degree, (6) Professional and/or Doctorate degree. Average of parents' education is calculated and reported.
Time Frame: Parent report, collected over 30 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | No Social Partner | Primary Parent | Experimenter
Number analyzed (Participants) | 67 | 65 | 56
scores on a scale | 4.5 (0.69) | 4.5 (0.83) | 4.5 (0.86)

24. Secondary Outcome: Caffeine or Nicotine Within 1 Hour of Testing. Potential Covariate
Description: Youth report on whether they consumed caffeine or nicotine in the 1-2 hours prior to the assessment. Coded as no=0, yes=1. Used as a potential covariate for heart rate and neuroendocrine measures.
Time Frame: Youth report, at start of 2 hour session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Social Partner | Primary Parent | Experimenter
Number analyzed (Participants) | 67 | 65 | 56
score on a scale | 0 (0) | 0 (0) | 0 (0)

25. Secondary Outcome: Granger Score
Description: The Granger score (ordinal, modeled continuously) is a score based on work by Doug Granger of medications that can affect activity of the HPA axis, weighted by significance of potential impact (Granger, Hibel, Fortunato, & Kapelewski, 2009). Each medication taken is given a score of 0, 1, or 2, and all medication scores for a participant is summed, resulting in scores from 0 to infinity. Lower scores are less likely to influence cortisol. Potential Covariate
Time Frame: Youth report at the beginning of the 2 hour session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Social Partner | Primary Parent | Experimenter
Number analyzed (Participants) | 66 | 63 | 56
score on a scale | 0.03 (0.25) | 0.19 (0.59) | 0.11 (0.41)

26. Secondary Outcome: Quality of Relationship With Primary Parent, BSV Positive Attachment Scale
Description: Network of Relationships Inventory (NRI) reported by youth for their primary parent on how much they experience various emotions or incidents (e.g. How much free time do you spend with this person?), reported on a 5-point scale: (1) Little or None, (2) Somewhat, (3) Very Much, (4) Extremely Much, (5) The Most. Mean scores calculated from all positive attachment items, range 1-5. Potential Covariate.
Time Frame: Youth report, collected over course of 30 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | No Social Partner | Primary Parent | Experimenter
Number analyzed (Participants) | 67 | 65 | 56
scores on a scale | 3.25 (0.69) | 3.12 (0.78) | 3.15 (0.74)

27. Secondary Outcome: Quality of Relationship With Close Friend, BSV Positive Attachment Scale
Description: Network of Relationships Inventory (NRI) reported by youth for their close friend on how much they experience various emotions or incidents (e.g. How much free time do you spend with this person?), reported on a 5-point scale: (1) Little or None, (2) Somewhat, (3) Very Much, (4) Extremely Much, (5) The Most. Mean scores calculated from all positive attachment items, ranging 1-5. Potential Covariate.
Time Frame: Youth reported, collected over course of 30 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | No Social Partner | Primary Parent | Experimenter
Number analyzed (Participants) | 67 | 65 | 56
scores on a scale | 3.36 (0.7) | 3.37 (0.75) | 3.43 (0.66)

ADVERSE EVENTS:
Time Frame: 1 DAY
Groups:
- No Social Partner: Participants will be randomly assigned to one of 3 conditions that differ by who is with them in the MRI scanner room: Primary Parent, Experimenter, No Social Partner.
  In this case, there was No Social Partner in the MRI room during the stressor.
- Primary Parent: Participants will be randomly assigned to one of 3 conditions that differ by who is with them in the MRI scanner room: Primary Parent, Experimenter, No Social Partner.
  In this case, the Primary Parent was in the MRI room during the stressor.
- Experimenter: Participants will be randomly assigned to one of 3 conditions that differ by who is with them in the MRI scanner room: Primary Parent, Experimenter, No Social Partner.
  In this case, the Experimenter was in the MRI room during the stressor.
Arm/Group | No Social Partner | Primary Parent | Experimenter
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/72 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/72 | 0/64
Other Adverse Events (participants affected / at risk) | 0/72 | 0/72 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/55/NCT04211155/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/55/NCT04211155/ICF_001.pdf